CLINICAL TRIAL: NCT03907566
Title: The Turkish Version of the Oropharyngeal Dysphagia Screening Test for Patients and Professionals
Brief Title: The Turkish Oropharyngeal Dysphagia Screening Test for Patients and Professionals
Status: Completed | Type: Observational
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, SELEN SEREL ARSLAN, Principal Investigator, Hacettepe University
Other Study IDs: Dysphagia screening
Record Dates: First submitted 2019-04-05; First posted 2019-04-09 (Actual); Last update posted 2024-01-05 (Actual); Status verified 2024-01

CONDITIONS: Swallowing Disorder
MeSH Terms: conditions — Deglutition Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Adult patients with swallowing disorders: Swallowing function will be evaluated with the Turkish Oropharyngeal Dysphagia Screening Test for Patients and Professionals, and Turkish version of the Eating Assessment Tool.
  Interventions: Other: The Turkish Oropharyngeal Dysphagia Screening Test for Patients and Professionals

INTERVENTIONS:
Other: The Turkish Oropharyngeal Dysphagia Screening Test for Patients and Professionals — Swallowing function will be evaluated by the Turkish Oropharyngeal Dysphagia Screening Test for Patients and Professionals

SUMMARY:
The purpose of this study is to test the reliability and validity of the The Turkish Oropharyngeal Dysphagia Screening Test for Patients and Professionals among adult patients with swallowing disorders.

DETAILED DESCRIPTION:
The purpose of this study is to test the reliability and validity of the The Turkish Oropharyngeal Dysphagia Screening Test for Patients and Professionals among adult patients with swallowing disorders.The internal consistency, test-retest reliability, and criterion validity of the instrument will be investigated. The internal consistency will be assessed using Cronbach's alpha. Intraclass correlation coefficient (ICC) value with 95 % confidence intervals will be calculated for test-retest reliability. The criterion validity of the scale will be determined by assessing the correlation between the The Turkish Oropharyngeal Dysphagia Screening Test for Patients and Professionals and Turkish Eating Assessment Tool.

ELIGIBILITY:
Inclusion Criteria:

* Willing to participate
* Having swallowing problems

Exclusion Criteria:

* Being under the age of 20 years, and above the age of 60 years
* Not willing to participate
* No swallowing problems

Ages: 20 Years to 60 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Study Population: Adult patients with swallowing concerns
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2019-05-01 (Actual); Primary Completion 2019-09-01 (Actual); Study Completion 2019-09-01 (Actual)

PRIMARY OUTCOMES:
The Turkish Oropharyngeal Dysphagia Screening Test for Patients and Professionals | 3 months
  This instrument is used to evaluate swallowing function. The test consists of 18 four points Likert-type items, organized assessing 3 scales: Safety, Efficacy, and Others. In most of the items, the Likert scale ranged from 1 = Never to 4 = Very often. The test score ranges from 18 (minimum) to 72 (maximum) points.

SECONDARY OUTCOMES:
The Turkish version of the Eating Assessment Tool-10 | 3 months
  The Turkish version of the Eating Assessment Tool-10 is a self-reporting instrument with 10 questions. Total score ranges between 0 to 40. Higher scores indicate worse swallowing function.

CONTACTS AND LOCATIONS:
Overall Officials: SELEN SEREL ARSLAN, Principal Investigator — Hacettepe University
Locations (1):
- Hacetttepe University, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No